CLINICAL TRIAL: NCT05975645
Title: A Phase Ib Clinical Study to Evaluate the Efficacy and Safety of TQB2618 Injection Combined With Penpulimab Injection and Anlotinib Hydrochloride Capsules as First-line Treatment for Advanced Hepatocellular Carcinoma.
Brief Title: A Clinical Study of TQB2618 Injection Combined With Penpulimab Injection and Anlotinib Hydrochloride Capsules for First-line Treatment of Advanced Hepatocellular Carcinoma (HCC).
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was closed due to business reasons. Closure was not prompted by any safety or efficacy concerns
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2618-AK105-Ib-04
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-06

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — penpulimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2618 injection +Penpulimab injection+ Anlotinib Hydrochloride Capsules (Experimental): Intravenous infusion of TQB2618 Injection 1200mg and Penpulimab Injection 200mg on 1st day, combining with Anlotinib capsules 10mg given orally in fasting conditions once daily in each 21-day cycle. (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21)
  Interventions: Drug: Penpulimab injection; Drug: TQB2618 injection; Drug: Anlotinib Hydrochloride Capsules

INTERVENTIONS:
Drug: Penpulimab injection — Penpulimab is an inhibitor of programmed cell death 1 (PD-1).
Drug: TQB2618 injection — TQB2618 injection is an inhibitor of T cell immunoglobulin and mucin domain-containing protein 3 (TIM-3).
Drug: Anlotinib Hydrochloride Capsules — Anlotinib hydrochloride is a muti-target tyrosine kinase inhibitor.

SUMMARY:
This is an open, single-arm, multi-center clinical study designed to evaluate the efficacy and safety of TQB2618 injection combined with penpulimab injection and Anlotinib Hydrochloride Capsules in patients with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old; Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1; Life expectancy ≥ 3 months.
* Patients with HCC diagnosed by histopathological or cytological examination or in line with clinical diagnostic criteria.
* No systematic treatment for advanced HCC has been received before.
* China liver cancer staging (CNLC)stage III or Barcelona Clinic Liver Cancer (BCLC) stage C, or CNLC stage II (BCLC B) subjects who are not suitable for local treatment and surgical treatment, or who are judged by researchers to be unable to benefit from local treatment and surgical treatment.
* Liver function score was good.
* Hepatitis B surface antigen (HBsAg) positive patients must meet hepatitis B virus deoxyribonucleic acid (HBV DNA) quantification < 10000 IU / ml (or 50000 copy/ml), and anti-HBV therapy should be given for at least 1 week before the first administration; investigator needs to determine that hepatitis C virus (HCV) infection is in a stable state.
* Patients after local treatment should be administered at least 4 weeks after the end of local treatment and have fully recovered from treatment toxicity and/or complications.
* Radiotherapy for bone metastases accompanied by clinical symptoms must be completed at least 2 weeks before the first administration.
* Has at least one measurable lesion.
* The Main organ function is normal.
* Men and women of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives, or condoms) during the study period and within 6 months after the end of the study. Serum human chorionic gonadotropin (HCG) test is not negative within 7 days before the first administration and must be non-lactating patients.
* Voluntary and signed informed consent, good compliance.

Exclusion Criteria:

* Combined disease and medical history :

  1. Other malignant tumors had appeared or were suffering from at the same time within 3 years before the first administration.
  2. Unrelieved toxic reactions higher than grade 1 due to any previous treatment.
  3. Major surgical treatment, obvious traumatic injury, or long-term unhealed wounds or fractures were received within 28 days before the first administration.
  4. Patients who had any bleeding or bleeding events ≥grade 3 within 8 weeks before the first administration, or had arterial/venous thrombosis events within 6 months before the first administration.
  5. There was a history of gastrointestinal bleeding within 6 months before the first administration; other conditions that may cause gastrointestinal bleeding or perforation.
  6. Patients with portal hypertension have a high risk of bleeding, or gastroscopy confirmed red sign or severe esophageal and gastric varices.
  7. Active pulmonary tuberculosis, history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonia, radiation pneumonitis requiring treatment, or active pneumonia with clinical symptoms.
  8. Have a history of mental drug abuse that cannot be withdrawn, or have a mental disorder.
  9. Patients who had previously received or planned to receive allogeneic bone marrow transplantation or solid organ transplantation within 6 months.
  10. Have a history of hepatic encephalopathy.
  11. Currently using or recently used aspirin (>325mg/day) or dipyridamole, ticlopidine, clopidogrel, and cilostazol treatment.
  12. Have any heavy and/or uncontrolled disease.
* Tumor-related, previous, and current treatment:

  1. Histopathology or cytology confirmed as fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, hepatobiliary cell carcinoma, mixed liver cancer, etc. Clinically considered as hepatobiliary mixed tumor.
  2. According to imaging examination, there was portal vein tumor thrombus involving the trunk; or inferior vena cava tumor thrombus or heart involvement.
  3. Subjects have been treated with immune checkpoint inhibitors such as programmed cell death protein 1 (PD-1), Programmed cell death 1 ligand 1(PD-L1), T cell immunoglobulin and mucin domain containing protein 3 (TIM-3), etc.
  4. Previously received any type of cellular immunotherapy.
  5. Has uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
  6. Suffering from spinal cord compression, cancerous meningitis, with symptoms of brain metastasis or symptoms control time less than 4 weeks.
* Study-related treatment:

  1. There was a history of attenuated live vaccine inoculation within 28 days before the first administration, or attenuated live vaccine inoculation was planned during the study period.
  2. Severe hypersensitivity reaction occurred after using macromolecular drugs.
  3. Those with multiple factors affecting the oral administration of drugs.
  4. Active autoimmune diseases requiring systemic treatment occurred within 2 years before the first administration.
  5. immunodeficiency, or Undergoing systemic glucocorticoid therapy or any other form of immunosuppressive therapy.
* Those who participated in and used other anti-tumor clinical trial drugs within 4 weeks before the first administration.
* According to the judgment of the investigators, some situations seriously endanger the safety of the subjects or affect the subjects to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years.
  Percentage of subjects achieving complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to two and a half years.
  OS is defined as the time from the first time the subject received treatment to death due to any cause.
Progress Free Survival (PFS) | Up to 2 years.
  The time from the first administration of the drug to disease progression or death (whichever occurs first).
Disease Control Rate (DCR) | Up to 2 years.
  Percentage of subjects achieving CR and PR and stable disease (SD) is greater than or equal to 4-6 weeks.
Duration of Response (DOR) | Up to 2 years.
  The time from the first assessment of the tumor's CR or PR to the disease's first progression or death from various causes.
Incidence of Anti-Drug antibody (ADA) | Before administration on the first day of the 1st, 2nd, 4th, and 8th cycles, 30 days and 90 days after the last administration. Each cycle is 21 days.
  The incidence of ADA after the administration of TQB2618.
Incidence of neutralizing antibodies (Nab) | Before administration on the first day of the 1st, 2nd, 4th, and 8th cycles, 30 days and 90 days after the last administration. Each cycle is 21 days.
  The incidence of Nab after the administration of TQB2618.
Incidence of adverse events (AEs) | Baseline up to 2 years.
  All adverse medical events that occur after the subject receives the investigational drug, evaluated according to the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0).
Severity of adverse events (AEs) | Baseline up to 2 years.
  All adverse medical events that occur after the subject receives the investigational drug, evaluated according to the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0).
Incidence of Serious adverse events (SAEs) | Baseline up to 2 years.
  It refers to adverse medical events such as death, life-threatening, permanent, or serious disability or loss of function, hospitalization or prolonged hospitalization, and congenital abnormalities or birth defects after the subject receives the experimental drug.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Gansu Wuwei Cancer Hospital, Wuwei, Gansu
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Affiliated hospital of zunyi medical university, Zunyi, Guizhou
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First People's Hospital of Shangqiu City, Shangqiu, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The six people's Hospital of Shenyang, Shenyang, Liaoning
  - Third Affiliated Hospital of Naval Medical University, Shanghai, Shanghai Municipality